CLINICAL TRIAL: NCT05660538
Title: A Phase 2, Randomized, Double-blind, Active-controlled, Dose-ranging, Parallel-design Study of the Efficacy and Safety of VX-548 in Subjects With Painful Diabetic Peripheral Neuropathy
Brief Title: Evaluation of Efficacy and Safety of VX-548 for Painful Diabetic Peripheral Neuropathy (DPN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX21-548-103
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Peripheral Neuropathy
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pregabalin (Active Comparator): Participants received Pregabalin 100 mg 3 times per day (tid) for 12 weeks
  Interventions: Drug: Pregabalin; Drug: Placebo (matched to SUZ)
- Suzetrigine (SUZ): Low Dose (Experimental): Participants received SUZ 23 mg tablet once daily (qd) for 12 weeks.
  Interventions: Drug: Suzetrigine; Drug: Placebo (matched to pregabalin)
- Suzetrigine (SUZ): Mid Dose (Experimental): Participants received SUZ 46 mg tablet qd for 12 weeks.
  Interventions: Drug: Suzetrigine; Drug: Placebo (matched to pregabalin)
- Suzetrigine (SUZ): High Dose (Experimental): Participants received SUZ 69 mg tablet qd for 12 weeks.
  Interventions: Drug: Suzetrigine; Drug: Placebo (matched to pregabalin)

INTERVENTIONS:
Drug: Suzetrigine — Tablets for oral administration.
  Other Names: VX-548; SUZ
  Arms: Suzetrigine (SUZ): High Dose; Suzetrigine (SUZ): Low Dose; Suzetrigine (SUZ): Mid Dose
Drug: Pregabalin — Capsules for oral administration.
  Arms: Pregabalin
Drug: Placebo (matched to SUZ) — Placebo matched to SUZ for oral administration.
  Arms: Pregabalin
Drug: Placebo (matched to pregabalin) — Placebo matched to pregabalin for oral administration.
  Arms: Suzetrigine (SUZ): High Dose; Suzetrigine (SUZ): Low Dose; Suzetrigine (SUZ): Mid Dose

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of VX-548 doses in treating Painful DPN.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of diabetes mellitus type 1 or type 2 with

  * Glycosylated hemoglobin A1c (HbA1c) ≤9%; and
  * Presence of bilateral pain in lower extremities due to DPN for at least 1 year

Key Exclusion Criteria:

* Painful neuropathy other than DPN
* History of cardiac dysrhythmias requiring anti-arrhythmia treatment(s)
* History of a clinical atherosclerotic event, such as myocardial infarction or stroke, within the past 12 months

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (50):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Synexus Clinical Research US - Birmingham, Birmingham, Alabama
  - Synexus Clinical Research US - Phoenix West, Phoenix, Arizona
  - Velocity Clinical Research - Banning, Banning, California
  - Long Beach Clinical Trials Services, Inc., Long Beach, California
  - University Clinical Investigators, Tustin, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - AMR Fort Myers (The Clinical Study Center), Fort Myers, Florida
  - Velocity Clinical Research - Hallandale Beach, Hallandale, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Accel Research Sites - Tampa, Largo, Florida
  - Accel Research Sites - Maitland, Maitland, Florida
  - Suncoast Research Associates, Miami, Florida
  - Synexus - Orlando, Orlando, Florida
  - Synexus - The Villages, The Villages, Florida
  - Accel Research Sites - Neurostudies, Decatur, Georgia
  - Velocity Clinical Research - Boise (Advanced Clinical Research), Meridian, Idaho
  - Healthcare Research Network - Chicago, Flossmoor, Illinois
  - Synexus Clinical Research - Evansville, Evansville, Indiana
  - AMR El Dorado, El Dorado, Kansas
  - AMR Newton, Newton, Kansas
  - AMR Wichita East, KS, Wichita, Kansas
  - Clinical Trials of America, LLC, Monroe, Louisiana
  - Brigham and Women's Hospital (BWH) - Translational Pain Research, Boston, Massachusetts
  - Boston Neuro Research Center, LLC, North Dartmouth, Massachusetts
  - Boston PainCare Center, Waltham, Massachusetts
  - Revival Research Institute, Dearborn, Michigan
  - StudyMetrix Research, LLC, City of Saint Peters, Missouri
  - Healthcare Research Network - Hazelwood, Hazelwood, Missouri
  - AMR Kansas City, Kansas City, Missouri
  - Synexus Clinical Research US - St. Louis, St Louis, Missouri
  - Synexus Clinical Research - Henderson, Henderson, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Synexus Clinical Research- New York, New York, New York
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Triad Clinical Trials, Greensboro, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Synexus - Cincinnati, Cincinnati, Ohio
  - Velocity Clinical Research - Cleveland, Cleveland, Ohio
  - Velocity Clinical Research - Medford, Medford, Oregon
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - Synexus Clinical Research- Anderson, Anderson, South Carolina
  - Clinical Trials of South Carolina - Charleston, Charleston, South Carolina
  - South Carolina Clinical Research, Orangeburg, South Carolina
  - Inquest Clinical Research, Baytown, Texas
  - Synexus - Dallas, Dallas, Texas
  - Diabetes & Glandular Disease Clinic, P.A, San Antonio, Texas
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Northwest Clinical Research Center (NWCRC), Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 194 participants were randomized in this study, out of which 192 participants received the study drug. Of these 192 participants, 19 participants from one of the sites were excluded due to lack of compliance with the study drug. Therefore, 173 participants are reported below for Baseline section and Efficacy outcomes and 192 participants are reported for Safety outcome and Adverse event section.
Period: Overall Study
Arm/Group | Pregabalin | Suzetrigine (SUZ): Low Dose | Suzetrigine (SUZ): Mid Dose | Suzetrigine (SUZ): High Dose
Started | 55 | 28 | 55 | 56
Safety Set (Safety set included all participants who received at least 1 dose of the study drug.) | 54 | 28 | 55 | 55
Modified Full Analysis Set (mFAS) (The mFAS is defined as all randomized participants who have received at least 1 dose of study drug and are not from Site 115.) | 49 | 24 | 50 | 50
Completed | 46 | 24 | 46 | 47
Not Completed | 9 | 4 | 9 | 9
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal of consent (not due to AE) | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Sponsor Decision | 1 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 1
Not completed — Randomized but did not receive study drug | 1 | 0 | 0 | 1
Not completed — Enrolled at clinical trial site excluded from mFAS due to lack of compliance with study drug | 5 | 4 | 5 | 5

BASELINE CHARACTERISTICS:
Population: Baseline data was analyzed based on the Modified Full Analysis Set (mFAS), defined as all randomized participants who have received at least 1 dose of study drug and are not from Site 115.
Groups:
- Pregabalin: Participants received Pregabalin 100 mg tid for 12 weeks.
- Suzetrigine (SUZ): Low Dose: Participants received SUZ 23 mg tablet qd for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Suzetrigine (SUZ): Low Dose | Suzetrigine (SUZ): Mid Dose | Suzetrigine (SUZ): High Dose | Total
Number analyzed (Participants) | 49 | 24 | 50 | 50 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (7.9) | 60.9 (6.6) | 61.7 (8.6) | 61.4 (8.8) | 61.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 12 | 22 | 21 | 77
  Male | 27 | 12 | 28 | 29 | 96
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9 | 4 | 22
  Not Hispanic or Latino | 42 | 22 | 41 | 46 | 151
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32 | 15 | 33 | 35 | 115
  Black or African American | 16 | 7 | 15 | 14 | 52
  Asian | 0 | 0 | 2 | 0 | 2
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 2
  Other | 0 | 1 | 0 | 0 | 1
  Multiracial | 0 | 1 | 0 | 0 | 1
Baseline Weekly Average Pain Intensity as Recorded on Numeric Pain Rating Scale (NPRS) [Mean (Standard Deviation); unit: units on a scale] — Population: Baseline weekly average pain intensity is defined as the average of non-missing pain intensity scores collected Days -7 to -1. Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0=no pain and 10=worst imaginable pain.Here "Number analyzed" signifies those participants who are evaluated for this specific baseline measure.
  units on a scale
    number analyzed (Participants) | 48 | 24 | 48 | 49 | 169
    (all) | 5.99 (1.27) | 5.70 (1.32) | 5.88 (0.97) | 5.83 (1.23) | 5.87 (1.18)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Average of Daily Pain Intensity on a Numeric Pain Rating Scale (NPRS)
Description: Change from baseline in the weekly mean of the daily Numeric Pain Rating Scale (NPRS) score assessing average pain intensity in the last 24 hours. Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain.
Time Frame: Baseline, At Week 12
Population: Modified Full Analysis Set (mFAS) included all randomized participants who have received at least 1 dose of study drug and are not from Site 115. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Suzetrigine (SUZ): High Dose: Participants received SUZ 69 mg tablet qd for 12 weeks.
  .
Arm/Group | Pregabalin | Suzetrigine (SUZ): Low Dose | Suzetrigine (SUZ): Mid Dose | Suzetrigine (SUZ): High Dose
Number analyzed (Participants) | 47 | 24 | 48 | 48
units on a scale | -2.09 [-2.65 to -1.52] | -2.18 [-2.94 to -1.41] | -2.11 [-2.67 to -1.55] | -2.26 [-2.82 to -1.70]

2. Secondary Outcome: Change From Baseline in the Weekly Average of the Daily Sleep Interference Scale (DSIS) Score
Description: Change from baseline in the weekly mean of the Daily Sleep Interference Scale (DSIS) score, which asks participants to describe how pain interfered with the participant's sleep. Response options for the DSIS range from 0 (none) to 10 (severe).
Time Frame: Baseline, At Week 12
Population: mFAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Pregabalin | Suzetrigine (SUZ): Low Dose | Suzetrigine (SUZ): Mid Dose | Suzetrigine (SUZ): High Dose
Number analyzed (Participants) | 47 | 24 | 49 | 47
units on a scale | -2.42 [-3.02 to -1.83] | -2.20 [-3.00 to -1.41] | -2.44 [-3.01 to -1.87] | -2.15 [-2.74 to -1.55]

3. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (≥) 30 Percent Reduction From Baseline in the Weekly Average of Daily Pain Intensity on the NPRS
Description: Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain.
  The percentage of participants with ≥30% reduction from baseline in the weekly average NPRS score at Week 12 was reported.
Time Frame: Baseline, At Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Suzetrigine (SUZ): Low Dose | Suzetrigine (SUZ): Mid Dose | Suzetrigine (SUZ): High Dose
Number analyzed (Participants) | 49 | 24 | 50 | 50
percentage of participants | 44.9 | 70.8 | 46.0 | 48.0

4. Secondary Outcome: Percentage of Participants With ≥50 Percent Reduction From Baseline in the Weekly Average of Daily Pain Intensity on the NPRS
Description: Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain.The percentage of participants with ≥50% reduction from baseline in the weekly average NPRS score at Week 12 was reported.
Time Frame: Baseline, At Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Suzetrigine (SUZ): Low Dose | Suzetrigine (SUZ): Mid Dose | Suzetrigine (SUZ): High Dose
Number analyzed (Participants) | 49 | 24 | 50 | 50
percentage of participants | 22.4 | 41.7 | 32.0 | 34.0

5. Secondary Outcome: Percentage of Participants With ≥70 Percent Reduction From Baseline in the Weekly Average of Daily Pain Intensity on the NPRS
Description: Pain intensity was recorded on 11-point NPRS, score range: 0 to 10, where 0= no pain and 10= worst imaginable pain.
  The percentage of participants with ≥70% reduction from baseline in the weekly average NPRS score at Week 12 was reported.
Time Frame: Baseline, At Week 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Suzetrigine (SUZ): Low Dose | Suzetrigine (SUZ): Mid Dose | Suzetrigine (SUZ): High Dose
Number analyzed (Participants) | 49 | 24 | 50 | 50
percentage of participants | 10.2 | 8.3 | 22.0 | 22.0

6. Secondary Outcome: Percentage of Participants Categorized as "Much Improved" or "Very Much Improved" on the Patient Global Impression of Change (PGIC) Assessment
Description: PGIC is an instrument that measures change in participants' overall status on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: Baseline, At Week 12
Population: mFAS.Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Suzetrigine (SUZ): Low Dose | Suzetrigine (SUZ): Mid Dose | Suzetrigine (SUZ): High Dose
Number analyzed (Participants) | 49 | 24 | 50 | 50
percentage of participants | 46.9 | 50.0 | 52.0 | 50.0

7. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 14
Population: Safety set included all participants who had received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin | Suzetrigine (SUZ): Low Dose | Suzetrigine (SUZ): Mid Dose | Suzetrigine (SUZ): High Dose
Number analyzed (Participants) | 54 | 28 | 55 | 55
Participants
  Participants with TEAEs | 20 | 14 | 21 | 31
  Participants with SAEs | 1 | 0 | 2 | 1

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 14
Description: Safety set included all participants who had received at least 1 dose of study drug.
Groups:
- Pregabalin: Participants received Pregabalin 100 mg 3 tid for 12 weeks.
Arm/Group | Pregabalin | Suzetrigine (SUZ): Low Dose | Suzetrigine (SUZ): Mid Dose | Suzetrigine (SUZ): High Dose
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/28 | 1/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/54 | 0/28 | 2/55 | 1/55
Other Adverse Events (participants affected / at risk) | 12/54 | 4/28 | 5/55 | 7/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=54) | Suzetrigine (SUZ): Low Dose (N=28) | Suzetrigine (SUZ): Mid Dose (N=55) | Suzetrigine (SUZ): High Dose (N=55)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=54) | Suzetrigine (SUZ): Low Dose (N=28) | Suzetrigine (SUZ): Mid Dose (N=55) | Suzetrigine (SUZ): High Dose (N=55)
Oedema peripheral (General disorders) | 3 | 1 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0 | 1 | 6
Weight increased (Investigations) | 4 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT05660538/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT05660538/SAP_001.pdf